CLINICAL TRIAL: NCT00979355
Title: Evaluation of Multi Purpose D-spect Camera for General Nuclear Scans
Brief Title: Study to Compare a Fast Gama Camera for Nuclear Imaging to Conventional Camera
Acronym: GP_D-Spect
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Spectrum Dynamics (Industry)
Responsible Party: Spectrum Dynamics, Spectrum Dynamics
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GP- DSpect_001
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Detect Pathalogical Lesions
Keywords: Whole body; SPECT

INTERVENTIONS:
Device: GP-D-SPECT — The D-SPECT system uses a solid-state detector, made of an alloy of Cadmium, Zinc, and Telluride, eliminating the need for thick crystals and large PMTs. As a result, the system is significantly miniaturized, and ergonomically optimized to both user and patient.

SUMMARY:
A feasibility trial to evaluate the usefulness of a high efficiency camera (D-SPECT) as an imaging modality for general nuclear medicine applications such as oncology.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is referred to nuclear medicine department for a SPECT scan.
2. Written informed consent is obtained by a study investigator.

Exclusion Criteria:

1. Patient pregnancy (known or suspected).
2. Lack of written informed consent
3. Prisoner status
4. Patient under age 18 or over 80 years old.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
A comparison of high efficiency camera images (D-SPECT) to a conventional camera (A-SPECT) with respect to the ability to detect pathological lesions. | 12 month

SECONDARY OUTCOMES:
A comparison of high efficiency camera images (D-SPECT) to a conventional camera (A-SPECT) with respect to image quality/resolution | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: MIGUEL GORENBERG, MD, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel